CLINICAL TRIAL: NCT06789263
Title: Clinical Study to Evaluate the Effect of a Collagen Hydrolysate on Postprandial Blood Glucose Profile, Gastric Emptying and GLP-1 Release in Normoglycemic and Prediabetic Subjects: Randomized, Double-blind, Placebo-controlled, Cross-over Design
Brief Title: Effect of a Collagen Hydrolysate on Postprandial Blood Glucose Profile, Gastric Emptying and GLP-1 Release in Normoglycemic and Prediabetic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rousselot BVBA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: BTS2127/24
Record Dates: First submitted 2025-01-15; First posted 2025-01-23 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Prediabetes; Normoglycemic
Keywords: glucose spikes; postprandial glucose; insulin response
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Collagen hydrolysate (Active Comparator): 30 min prior to the mixed meal test
  Interventions: Dietary Supplement: Collagen hydrolyzed peptides
- Placebo (Placebo Comparator): Flavoured water
  Interventions: Other: Placebo
- Collagen hydrolysate II (Other): together with the mixed meal test
  Interventions: Dietary Supplement: Collagen hydrolyzed peptides

INTERVENTIONS:
Dietary Supplement: Collagen hydrolyzed peptides — Dissolved in flavoured water, single dose, 10 g
  Arms: Collagen hydrolysate; Collagen hydrolysate II
Other: Placebo — Single dose
  Arms: Placebo

SUMMARY:
Aim of the study is to investigate the postprandial response on blood glucose, insulin, C-peptide, incretin response and gastric emptying after intake of collagen hydrolysate compared to placebo in normoglycemic and in prediabetic participants. This will be investigated in a cross-over randomized double-blind placebo controlled study design.

In an exploratory part II, timing of intake of collagen hydrolysate in relation to the mixed meal will be investigated in a subgroup of 50% of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Prediabetic subjects: Male and female subjects with prediabetic HbA1c values between 5.7% and 6.4% and/or fasting glucose ≥ 100 mg/dL and ≤ 125 mg/dL (in venous plasma) (twice confirmed at two independent days if HbA1c is < 5.7%) or Healthy normoglycemic subjects: fasting glucose <100 mg/dL and HbA1c is < 5.7%
* Age: 18-70 years
* Body mass index 19-35 kg/m2
* Current Non-smoker
* Signed informed consent form
* No changes in food habits or physical activity 3 months prior to screening and during the study
* If applicable, stable intake of chronic medication of at least 4 weeks

Exclusion Criteria:

* Subjects with diagnosed Type 2 Diabetes mellitus with medical treatment
* Presence of disease or drug(s) influencing digestion (incl. recent intake of antibiotics) and absorption of nutrients
* Intake of medications known to affect glucose tolerance, e.g., diabetic medication, SGLT-2 inhibitors, GLP-1 receptor agonists, steroids, protease inhibitors or antipsychotics
* Chronic intake of substances affecting blood coagulation (e.g. acetylic acid (100 mg as standard prophylactic treatment allowed when dose is stable 1 month prior to screening), anticoagulants, diuretics, thiazides (diuretics and thiazides allowed e.g. for hypertension treatment when dose is stable 1 month prior to screening), which in the Investigator's opinion would impact patient safety
* Severe liver or renal disease or laboratory evidence of hepatic dysfunction (i.e. alkaline phosphatase, ALT, AST >3 x ULN)
* Known inflammatory or malignant gastrointestinal diseases (i.e. colitis ulcerosa, Morbus Crohn, celiac disease, malignant diseases e.g. colon-cancer, rectum cancer, pancreatitis)
* Subjects who use an implanted or portable electro-mechanical medical device such as a cardiac pacemaker or infusion pump.
* Planned MRI during or 4 weeks after the study.
* Subjects overweighed with abdominal diameter >140 cm
* Clinically relevant findings as established by medical history, physical examination, clinical laboratory and/or vital signs
* Major medical or surgical event requiring hospitalization within the previous 3 months
* Intake of food supplements known to affect glucose tolerance, e.g., cinnamon capsules, conjugated linoleic acids
* Drug-, alcohol- and medication abuses
* Pregnant or breast-feeding women
* Weight loss intervention or recent body weight change >5 kg during the last 3 months
* Blood donation within 4 weeks prior to Screeningor plan to donate blood during the study
* Anticipating any planned changes in lifestyle for the duration of the study
* Participation in another clinical intervention study within the last 4 weeks and concurrent participation in another intervention clinical study
* Subjects considered inappropriate for the study by investigators, including subjects who are unable or unwilling to show compliance with the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Glucose iAUC | 0-180 minutes postprandially
  Area under the curve (AUC) calculated as the incremental area under the blood glucose response curve, ignoring the area beneath the fasting concentration: Glucose-iAUC(0-180minutes)

SECONDARY OUTCOMES:
Glucose Cmax | 0-180 minutes postprandially
  Maximum blood glucose concentration (Cmax)
Delta Cmax | 0-180 minutes postprandially
  Maximum increase of blood glucose concentration
Tmax | 0-180 minutes postprandially
  Time to reach maximum blood glucose concentration (Tmax)
Fasting glucose | -30 minutes and 0 minutes prior mixed meal
  Fasting glucose
Glucose | 120 minutes
  Blood glucose concentration after mixed meal
Fasting insulin | -30 minutes and 0 minutes prior to mixed meal
  Fasting insulin
Insulin iAUC | 0-180 minutes postprandially
  Area under the curve calculated as the incremental area under the insulin curve
Fasting C-peptide | -30 minutes and 0 minutes prior mixed meal
  Fasting C-peptide
C-peptide iAUC | 0-180 minutes postprandially
  Area under the curve calculated as the incremental area under the C-peptide curve
GLP-1 iAUC | 0-120 minutes postprandially
  Incretin response (Glucagon-like Peptide-1)
Fasting GLP-1 | -30 minutes and 0 minutes prior mixed meal
  Fasting GLP-1
Matsuda-Index | 0-120 minutes postprandially
  Determination of Insulin sensitivity
Gastric emptying | 0-6 hours postprandially
  Time for gastric emptying
Satiety assessment | 0-240 minutes postprandially
  Visual analog scale (VAS) Scale (0: not at all 100: extremely)

OTHER OUTCOMES:
Gastrointestinal hormones | 0-120 minutes postprandially
  Glucose-dependent insulinotropic polypeptide (GIP)

CONTACTS AND LOCATIONS:
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: No